CLINICAL TRIAL: NCT00000173
Title: A Randomized, Double-Blind, Placebo-Controlled Trial of Vitamin E and Donepezil HCL (Aricept) to Delay Clinical Progression From Mild Cognitive Impairment (MCI) to Alzheimer's Disease (AD)
Brief Title: Memory Impairment Study (Mild Cognitive Impairment Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: Alzheimer's Disease Cooperative Study (ADCS) (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IA0011; 3U01AG010483-08S2 (NIH)
Record Dates: First submitted 1999-10-29; First posted 1999-11-01 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2009-06

CONDITIONS: Alzheimer Disease
Keywords: Mild cognitive impairment; Alzheimer's disease; Memory; Donepezil; Vitamin E; Antioxidants; Cholinergic agents; Cholinesterase inhibitors
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — Donepezil; Vitamin E

INTERVENTIONS:
Drug: Donepezil
Drug: Vitamin E

SUMMARY:
The National Institute on Aging (NIA) is launching a nationwide treatment study targeting individuals with mild cognitive impairment (MCI), a condition characterized by a memory deficit, but not dementia. An NIA-funded study recently confirmed that MCI is different from both dementia and normal age-related changes in memory. Accurate and early evaluation and treatment of MCI individuals might prevent further cognitive decline, including development of Alzheimer's disease (AD).

The Memory Impairment Study is the first such AD prevention clinical trial carried out by NIH, and will be conducted at 65-80 medical research institutions located in the United States and Canada. This study will test the usefulness of two drugs to slow or stop the conversion from MCI to AD. The trial will evaluate placebo, vitamin E, and donepezil, an investigational agent approved by the Food and Drug Administration for another use. Vitamin E (alpha-tocopherol) is thought to have antioxidant properties, and was shown in a 1997 study to delay important dementia milestones, such as patients' institutionalization or progression to severe dementia, by about seven months.

DETAILED DESCRIPTION:
This clinical trial will be a multicenter, randomized, double-blind, placebo- controlled, parallel-group study of vitamin E and donepezil in 720 subjects with mild cognitive impairment (MCI). Subjects will be randomized to one of three treatment groups (240 subjects per treatment group): 1) Placebo vitamin E and placebo donepezil plus a multivitamin daily. 2) Vitamin E (2,000 I) and placebo donepezil plus a multivitamin daily.3) Donepezil (10 mg) and placebo vitamin E plus a multivitamin daily.

The study will be conducted over three years, with clinical evaluations every 3 months for the first 6 months and then every 6 months. Subjects randomized to donepezil will start a dose of 5 mg daily. Donepezil will be increased to 10 mg after six weeks. Subjects randomized to vitamin E will start at 1,000 I daily. The dose of Vitamin E will be increased to 2,000 I after six weeks. There will be a 12-month recruitment period. The primary endpoint will be time to development of Probable or Possible AD according to NINCDS-ADRDA criteria. Upon determination of a clinical diagnosis of AD, documentation will be sent to the ADCS Coordinating Center and forwarded to the Central Review Committee for verification. Upon verification, of conversion to diagnosis of AD, subjects will stop taking the donepezil study medication or its corresponding placebo, without breaking the blind, and will be offered open label donepezil at a scheduled visit one month after the prior diagnostic visit. Donepezil will be offered to subjects who convert to AD until the subject completes three years from the baseline visit. Based on an estimated incidence of AD of 15% per year, the study has 85% power to detect a 33% or greater reduction in conversion to AD over 3 years. Secondary outcome measures will include change on the Alzheimer's Disease Assessment Scale (ADAS-COG), the Neuropsychological Battery, the Mini-Mental State Exam (MMSE), Clinical Dementia Rating Scale (CDR), the Global Deterioration Scale (GDS), ADCS- Activities of Daily Living Inventory (ADCS-ADL), a Pharmacoeconomics scale, and a Quality of Life scale. Compliance will be monitored through the measurement of alpha-tocopherol levels and pill counts at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Memory complaints and memory difficulties which are verified by an informant.
* Abnormal memory function documented by scoring below the education adjusted cutoff on the Logical Memory II subscale (Delayed Paragraph Recall) from the Wechsler Memory Scale - Revised (the maximum score is 25): a) less than or equal to 8 for 16 or more years of education, b) less than or equal to 4 for 8-15 years of education, c) less than or equal to 2 for 0-7 years of education.
* Mini-Mental Exam score between 24 and 30 (inclusive) (Exceptions may be made for subjects with less than 8 years of education at the discretion of the project director.).
* Clinical Dementia Rating = 0.5. Memory Box score must be at least 0.5.
* General cognition and functional performance sufficiently preserved such that a diagnosis of Alzheimer's disease cannot be made by the site physician at the time of the screening visit.
* No significant cerebrovascular disease: Modified Hachinski score of less than or equal to 4.
* Age between 55 and 90 (inclusive).
* Permitted medications stable for at least 1 month prior to screening. In particular: a) Subjects may take stable doses of antidepressants lacking significant anticholinergic side effects (if they are not currently depressed and do not have a history of major depression within the past 2 years). b) Estrogen replacement therapy is permissible. c) Ginkgo biloba is permissible, but discouraged.
* Hamilton Depression rating scale score of less than or equal to 12 on the 17-item scale.
* Informant is available who has frequent contact with the subject (e.g. an average of 10 hours per week or more), agrees to monitor administration of study drug, observe for adverse events, and accompany the subject to all clinic visits for the duration of the protocol.
* CT or MRI scans within 12 months prior to screening without evidence of infection, infarction, or other focal lesions and without clinical symptoms suggestive of intervening neurological disease. A lacune in a non-critical brain area which is not believed to contribute to the subject's cognitive impairment is permissible.
* Adequate visual and auditory acuity to allow neuropsychological testing.
* Good general health with no additional diseases expected to interfere with the study.
* Normal B12, RPR, and Thyroid Function Tests or without any clinically significant abnormalities that would be expected to interfere with the study.
* ECG without clinically significant abnormalities that would be expected to interfere with the study.
* Subject is not pregnant, lactating, or of childbearing potential (i.e. women must be two years post-menopausal or surgically sterile).
* Agreement not to take other vitamin supplements (including Vitamin E), multivitamins, other than those provided by the study.

Exclusion Criteria:

* Any significant neurologic disease other than suspected incipient Alzheimer's disease, such as Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities.
* Major depression or another major psychiatric disorder as described in DSM IV within the past 2 years.
* Psychotic features, agitation or behavioral problems within the last 3 months which could lead to difficulty complying with the protocol.
* History of alcohol or substance abuse or dependence within the past 2 years (DSM IV criteria).
* History of schizophrenia (DSM IV criteria).
* Any significant systemic illness or unstable medical condition which could lead to difficulty complying with the protocol including: a) History of systemic cancer within the last 5 years (non-metastatic skin cancers are acceptable). b) History of myocardial infarction within the past year or unstable or severe cardiovascular disease including angina or CHF with symptoms at rest. c) Clinically significant obstructive pulmonary disease or asthma. d) Clinically significant and unstable gastrointestinal disorder such as ulcer disease or a history of active or occult gastrointestinal bleeding within two years. e) Clinically significant laboratory test abnormalities on the battery of screening tests (hematology, prothrombin time, chemistry, urinalysis, ECG). f) Insulin-requiring diabetes or uncontrolled diabetes mellitus. g) Uncontrolled hypertension (systolic BP greater than 170 or diastolic greater than 100). h) History of clinically significant liver disease, coagulopathy, or vitamin K deficiency within the past 2 years.
* Medications a) Use of centrally active beta-blockers, narcotics, methyldopa and clonidine within 4 weeks prior to screening. b) Use of anti-Parkinsonian medications (e.g. Sinemet, amantadine, bromocriptine, pergolide and selegiline) within 2 months prior to screening. c) Use of neuroleptics or narcotic analgesics within 4 weeks prior to screening. d) Use of long-acting benzodiazepines or barbituates within 4 weeks prior to screening. e) Use of short-acting anxiolytics or sedative hypnotics more frequently than 2 times per week within 4 weeks prior to screening (note: sedative agents should not be used within 72 hours of screening).

  f) Initiation or change in dose of an antidepressant lacking significant cholinergic side effects within the 4 weeks prior to screening (use of stable doses of antidepressants for at least 4 weeks prior to screening is acceptable). g) Use of systemic corticosteroids within 3 months prior to screening. h) Medications with significant cholinergic or anticholinergic side effects (e.g. pyridostigmine, tricyclic antidepressants, meclizine, and oxybutynin) within 4 weeks prior to screening. i) Use of anti-convulsants (e.g. Phenytoin, Phenobarbital, Carbamazepine) within 2 months prior to screening. j) Use of warfarin (Coumadin) within 4 weeks prior to screening.
* Vitamin Supplements a) Use of vitamin supplements other than standard multivitamin included as part of the treatment intervention used in this protocol within 2 weeks prior to screening.
* Any prior use of any FDA approved medications for the treatment of Alzheimer's disease (e.g. tacrine, donepezil, or other newly approved medications).
* Use of any investigational drugs within 30 days or 5 half-lives, whichever is longer, prior to screening.
* Subjects who, in the investigator's opinion, will not comply with study procedures.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-03; Primary Completion 2004-01 (Actual); Study Completion 2004-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leon Thal, MD, Principal Investigator — Alzheimer's Disease Cooperative Study
Locations (72):
- United States (63):
  - Barrow Neurological Group, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - UC Irvine Institute for Brain Aging and Dementia, Irvine, California
  - University of Southern California, Los Angeles, California
  - University of California, Los Angeles, Los Angeles, California
  - East Bay Institute, Martinez, California
  - Sutter Institute for Medical Research, Sacramento, California
  - Affiliated Research Instiute, San Diego, California
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Yale University, New Haven, Connecticut
  - Baumel-Eisner Neuromedical Institute, Boca Raton, Boca Raton, Florida
  - Baumel-Eisner Neuromedical Institute, Ft. Lauderdale, Fort Lauderdale, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Wein Center, Miami Beach, Florida
  - Baumel-Eisner Neuromedical Institute, MiamiBeach, Miami Beach, Florida
  - University of Miami, Port Charlotte, Florida
  - University of South Florida, Tampa, Florida
  - Premiere Research Institute, West Palm Beach, Florida
  - Emory University, Atlanta, Georgia
  - Augusta VA Medical Center, Augusta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush Presbyterian St. Luke's Medical Center, Chicago, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - University of Nevada, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Memory Disorders Institute, Lakehurst, New Jersey
  - Princeton Biomedical Research, PA, Princeton, New Jersey
  - ClinSearch, Inc., Summit, New Jersey
  - Princeton Biomedical - Toms River, Toms River, New Jersey
  - Alzheimer's Research Corp., West Long Branch, New Jersey
  - Univ. of New Mexico, Albuquerque, New Mexico
  - Maimonides Medical Center, Brooklyn, New York
  - NYU Medical Center, New York, New York
  - Mount Sinai Medical Center, New York, New York
  - Columbia University, New York, New York
  - Nathan S. Kline Institute for Psychiatric Research, Orangeburg, New York
  - University of Rochester, Rochester, New York
  - SUNY Stony Brook, Stony Brook, New York
  - Burke Medical Research Institute, White Plains, New York
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - MCP Hahnemann, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Brown University, Pawtucket, Rhode Island
  - Medical University of South Carolina, North Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Southwestern Vermont Medical Center, Bennington, Vermont
  - Clinical Neuroscience Research Unit, Burlington, Vermont
  - University of Washington, Seattle, Washington
  - Marshfield Clinic, Marshfield, Wisconsin
- Canada (9):
  - University of Calgary, Calgary, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - Fredericton Medical Clinic, Fredericton, New Brunswick
  - Geriatric Medicine Research Group, Halifax, Nova Scotia
  - St. Joseph's Health Center, London, Ontario
  - Elizabeth Bruyere Centre, Ottawa, Ontario
  - Sunnybrook Health Science Center, Toronto, Ontario
  - Jewish General Hospital Memory Clinic, Montreal, Quebec
  - McGill Centre for Studies in Aging, Verdun, Quebec

REFERENCES:
- [Background] Rogers SL, Farlow MR, Doody RS, Mohs R, Friedhoff LT. A 24-week, double-blind, placebo-controlled trial of donepezil in patients with Alzheimer's disease. Donepezil Study Group. Neurology. 1998 Jan;50(1):136-45. doi: 10.1212/wnl.50.1.136. PMID 9443470
- [Background] Petersen RC, Smith GE, Waring SC, Ivnik RJ, Kokmen E, Tangelos EG. Aging, memory, and mild cognitive impairment. Int Psychogeriatr. 1997;9 Suppl 1:65-9. doi: 10.1017/s1041610297004717. PMID 9447429
- [Background] Rubin EH, Morris JC, Grant EA, Vendegna T. Very mild senile dementia of the Alzheimer type. I. Clinical assessment. Arch Neurol. 1989 Apr;46(4):379-82. doi: 10.1001/archneur.1989.00520400033016. PMID 2650663
- [Result] Grundman M, Petersen RC, Ferris SH, Thomas RG, Aisen PS, Bennett DA, Foster NL, Jack CR Jr, Galasko DR, Doody R, Kaye J, Sano M, Mohs R, Gauthier S, Kim HT, Jin S, Schultz AN, Schafer K, Mulnard R, van Dyck CH, Mintzer J, Zamrini EY, Cahn-Weiner D, Thal LJ; Alzheimer's Disease Cooperative Study. Mild cognitive impairment can be distinguished from Alzheimer disease and normal aging for clinical trials. Arch Neurol. 2004 Jan;61(1):59-66. doi: 10.1001/archneur.61.1.59. PMID 14732621
- [Derived] Potashman M, Pang M, Tahir M, Shahraz S, Dichter S, Perneczky R, Nolte S. Psychometric properties of the Alzheimer's Disease Cooperative Study - Activities of Daily Living for Mild Cognitive Impairment (ADCS-MCI-ADL) scale: a post hoc analysis of the ADCS ADC-008 trial. BMC Geriatr. 2023 Mar 6;23(1):124. doi: 10.1186/s12877-022-03527-0. PMID 36879199
- [Derived] Lansdall CJ, McDougall F, Butler LM, Delmar P, Pross N, Qin S, McLeod L, Zhou X, Kerchner GA, Doody RS. Establishing Clinically Meaningful Change on Outcome Assessments Frequently Used in Trials of Mild Cognitive Impairment Due to Alzheimer's Disease. J Prev Alzheimers Dis. 2023;10(1):9-18. doi: 10.14283/jpad.2022.102. PMID 36641605
- [Derived] Donohue MC, Langford O, Insel PS, van Dyck CH, Petersen RC, Craft S, Sethuraman G, Raman R, Aisen PS; Alzheimer's Disease Neuroimaging Initiative. Natural cubic splines for the analysis of Alzheimer's clinical trials. Pharm Stat. 2023 May-Jun;22(3):508-519. doi: 10.1002/pst.2285. Epub 2023 Jan 10. PMID 36627206
- [Derived] Oxtoby NP, Shand C, Cash DM, Alexander DC, Barkhof F. Targeted Screening for Alzheimer's Disease Clinical Trials Using Data-Driven Disease Progression Models. Front Artif Intell. 2022 May 26;5:660581. doi: 10.3389/frai.2022.660581. eCollection 2022. PMID 35719690
- [Derived] DeCarli C, Frisoni GB, Clark CM, Harvey D, Grundman M, Petersen RC, Thal LJ, Jin S, Jack CR Jr, Scheltens P; Alzheimer's Disease Cooperative Study Group. Qualitative estimates of medial temporal atrophy as a predictor of progression from mild cognitive impairment to dementia. Arch Neurol. 2007 Jan;64(1):108-15. doi: 10.1001/archneur.64.1.108. PMID 17210817
- See also: More information about the study from the Alzheimer's Disease Cooperative Study site at the University of California at San Diego. — http://adcs.ucsd.edu
- See also: The Alzheimer's Disease Education and Referral (ADEAR) Center is a service of the National Institute on Aging. — http://www.alzheimers.org